CLINICAL TRIAL: NCT05033821
Title: A Library-based Prevention Intervention for Adolescents Affected by Parental Drug Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: K01
Record Dates: First submitted 2021-07-30; First posted 2021-09-05 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Substance Use; Sexual Behavior; Adolescent Behavior
Keywords: substance use prevention; adolescent health; selective intervention; community-based research; parental drug use
MeSH Terms: conditions — Substance-Related Disorders; Sexual Behavior; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants who receive the FOY+ImPACT intervention
  Interventions: Behavioral: Adapted FOY+ImPACT
- Control (No Intervention): Participants who receive standard library programing, but not the FOY+ImPACT intervention.

INTERVENTIONS:
Behavioral: Adapted FOY+ImPACT — The Adapted FOY+IMPACT is a selective, group-level intervention designed to prevent sexual risk-taking and substance use among adolescents affected by parental drug use. There are eight sessions for youth (FOY) and one session with youth and adults (ImPACT).
  Arms: Intervention

SUMMARY:
This study's goal is to partner with public libraries to prevent substance use and sexual risk-taking among urban African American adolescents (ages 13-16) affected by parental drug use. An existing universal evidence-based intervention (Focus on Youth with Informed Parents and Children Together, abbreviated as FOY+ImPACT) will be adapted for adolescents affected by parental drug use and delivered in libraries. FOY+ImPACT is a skill-building intervention aimed at preventing substance use and sexual risk-taking among high-risk African American youth. The investigative team will conduct a pilot study to assess the feasibility and initial efficacy of a library-based prevention intervention for adolescents affected by drug use. Participants will be Black adolescents (13-16 years old) affected by parental drug use (N=120). Adolescents will be randomized by partner organization to receive the intervention virtually. Pre, Post and 3-month follow-up data will be collected using computerized surveys. Primary outcomes will be substance use (i.e., marijuana and alcohol use, two of the most common drugs for this age group) and sexual risk behaviors (i.e., initiation of sex and frequency of unprotected sex).

DETAILED DESCRIPTION:
With nearly 17,000 public libraries nationwide and four million visits each day, libraries have extensive population reach. Libraries are an ideal partner because they are stable, safe, accessible, confidential community spaces with a low barrier to entry and non-judgmental staff. This study's goal is to partner with public libraries to prevent substance use and sexual risk-taking among urban African American adolescents (ages 13-16) affected by parental drug use. An existing universal evidence-based intervention (Focus on Youth with Informed Parents and Children Together, abbreviated as FOY+ImPACT) will be adapted for adolescents affected by parental drug use and delivered in libraries. FOY+ImPACT is a skill-building intervention aimed at preventing substance use and sexual risk-taking among high-risk African American youth.

For this study, a 'parent with a history of drug use' is defined as a biological parent who abused an illicit drug for longer than 1 month in the past 2 years. This group includes parents in recent recovery and those enrolled in substance abuse treatment programs. Many youth affected by parental drug use live with someone who does not use drugs, extended family members, or are in the care of social services. Thus, primary caregivers will be eligible to participate in the absence of a biological parent. A 'primary caregiver', is defined as a person who regularly provides care for a child that is not their birth child.

The investigative team will conduct a pilot study to assess the feasibility and initial efficacy of a library-based prevention intervention for adolescents affected by drug use. Participants will be Black adolescents (13-16 years old) affected by parental drug use (N=120). Adolescents will be randomized by partner organization to receive the intervention virtually. Pre, Post and 3-month follow-up data will be collected using computerized surveys. Primary outcomes will be substance use (i.e., marijuana and alcohol use, two of the most common drugs for this age group) and sexual risk behaviors (i.e., initiation of sex and frequency of unprotected sex).

ELIGIBILITY:
Inclusion Criteria:

* Black/African American
* 13-16 years old
* have a caregiver with a history of drug use
* English-speaking

Exclusion Criteria:

-

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Change in youth substance use based on Youth Risk Behavior Surveillance Survey | baseline, post intervention and 3 months
  The Youth Risk Behavior Surveillance Survey (YRBS) monitors six categories of health-related behaviors that contribute to the leading causes of death and disability among youth and adults, including alcohol and other drug use. The survey asks about frequency current use (i.e., number of days in the past 30 days) of alcohol and other drugs. Responses for each substance can be "0 days", "1 or 2 days", "3 to 5 days", "6 to 9 days", "10 to 19 days", "20 to 29 days", or "all 30 days".
2. Change in youth sexual risk-taking based on Youth Risk Behavior Surveillance Survey | baseline, post intervention and 3 months
  The Youth Risk Behavior Surveillance Survey (YRBS) monitors six categories of health-related behaviors that contribute to the leading causes of death and disability among youth and adults, including Sexual behaviors related to unintended pregnancy and sexually transmitted diseases, including HIV infection. The survey asks about initiation of sex and frequency of unprotected sex. Responses for sexual initiation are "yes" or "no". Responses for other contraceptive use at last sex are "I have never had sexual intercourse ", "No method was used to prevent pregnancy", "birth control pills", "Condoms", "An intrauterine device (IUD, such as Mirena or ParaGard) or implant (such as Implanon or Nexplanon)", "A shot (such as Depo-Provera)", "patch (such as Ortho Evra), or birth control ring (such as NuvaRing)", "Withdrawal or some other method", and "Not sure".

CONTACTS AND LOCATIONS:
Overall Officials: Terrinieka Powell, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Powell TW, Willis K, Smith B, Lewis Q, Offiong A. "Don't Close the Door on Them": Recruiting and retaining vulnerable Black adolescents in prevention research. J Community Psychol. 2021 Jul;49(5):994-1009. doi: 10.1002/jcop.22584. Epub 2021 May 3. PMID 33937999
- [Background] Offiong A, Powell TW, Lewis Q, Smith B, Prioleau M. "I missed open arms": The Need for Connectedness among Black Youth Affected by Parental Drug Use. Child Youth Serv Rev. 2020 Jul;114:105072. doi: 10.1016/j.childyouth.2020.105072. Epub 2020 May 8. PMID 32606485
- [Background] Lewis QJ, Smith BD, Offiong A, Prioleau M, Powell TW. When a house is never a home: Housing instability among youth affected by parental drug abuse. Child Abuse Negl. 2021 Aug;118:105131. doi: 10.1016/j.chiabu.2021.105131. Epub 2021 Jun 9. PMID 34118586
- [Derived] Powell T, Smith BD, Moser N, Kachingwe O, Lewis Wallace Q, Offiong A, Hwang A, Davie E, LoVette A. Adapting a Sexual Health Intervention for Adolescents Exposed to Adversity: Feasibility Study. JMIR Form Res. 2026 Jan 5;10:e72782. doi: 10.2196/72782. PMID 41490399
- See also: Related Info — http://www.researchbypowell.com